CLINICAL TRIAL: NCT05436132
Title: The Effects of Virtual Reality and Augmented Reality (VR/AR) Educational Module on Oral Care Practices for Home Care Worker
Brief Title: VR/AR Educational Module on Oral Care Practices for Home Care Worker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KMUHIRB- F(I)-20200098
Record Dates: First submitted 2022-06-21; First posted 2022-06-28 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2022-06

CONDITIONS: Virtual Reality; Augmented Reality; Oral Care Performance
Keywords: Virtual reality; Augmented reality; Oral Care Performance; home care worker; elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR/AR group (Experimental): Home care workers (HCW)HCWs in the VR/AR group received 2.5 hours of VR and AR training. VR offered learners the standard oral care procedures under different physical and oral health conditions in elderly people and AR simulation training for the manual Bass brushing technique.
  Interventions: Behavioral: VR and AR oral healthcare curriculum training
- Control group (Placebo Comparator): The home care workers in the control group received 2.5 hours of traditional teaching methods for oral care.
  Interventions: Behavioral: traditional teaching methods oral healthcare curriculum

INTERVENTIONS:
Behavioral: VR and AR oral healthcare curriculum training — HCWs in the VR/AR group received 2.5 hours VR and AR oral healthcare curriculum training. VR oral care training system was training the standard oral healthcare procedure for different physical and oral conditions in elderly people.AR oral care training system was training for the manual Bass brushing technique.
  Arms: VR/AR group
Behavioral: traditional teaching methods oral healthcare curriculum — HCWs in the control group received 2.5 hours traditional teaching methods of oral healthcare curriculum training.
  Arms: Control group

SUMMARY:
This study is to evaluate the effect of the elderly oral care knowledge, attitude ,self-efficacy ,oral care behavior between the home care workers(HCW) in VR(Virtual reality)/AR(Augmented reality)group and control group after intervention. Home care workers will be randomly assigned to the VR/AR group and the control group. Home care workers in the VR/AR group will use VR to learned about the oral care methods and processes in the different case. AR allows HCWs to actually operate cleaning teeth. The home care workers in the control group used traditional teaching methods for oral care. Baseline and follow-up survey were used to collect the data in oral care knowledge, attitude ,self-efficacy ,oral care behavior.

DETAILED DESCRIPTION:
A randomized experimental design was used. Home care workers (HCWs) in the VR/AR group received 2.5 hours of VR(Virtual reality) and AR(Augmented reality) training. VR offered learners the standard oral care procedures under different physical and oral health conditions in elderly people and AR simulation training for the manual Bass brushing technique. The home care workers in the control group used traditional teaching methods for oral care. A self-administered questionnaire was used to collect data regarding oral care-related knowledge, attitude, self-efficacy, intention to assist in oral care behavior and behavior before and after the intervention, 3-month follow-up and 6-month follow-up. All participants finished the self-administered questionnaire within 10-15 minutes and handed it to researchers at VR/AR oral care training center in Kaohsiung Medical University.Generalized estimating equations (GEEs) was used to analyze the differences between pre-test, post-test and follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* certificated home care workers in Taiwan.

Exclusion Criteria:

* aged above 65 were excluded.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
oral care behavior | Change from 3-month follow-up to 6-month follow-up. After two groups HCWs received the intervention, 3 months and 6 months HCWs would received follow-up questionnaire to finish the measurement.
  Eight statements were used to evaluate the behavior in assisting in oral care behavior Item including that" I take the initiative to assist the elderly to perform oral care ." All response was coded as zero (not) or one (yes).

SECONDARY OUTCOMES:
Oral care-related knowledge | After randomization, HCWs would receive pre-test before intervention and post-test after intervention immediately. The follow-up questionnaire to measure at 3 months and 6 months after intervention.
  Ten statements were used to assess oral care-related knowledge. Item including that" Fluoride toothpaste for adults should have a fluoride content above 1000 ppm." A score of 0 (incorrect) and 1 (correct) was used for each statement. The total score ranged was 0-10.
Attitude toward oral care | After randomization, HCWs would receive pre-test before intervention and post-test after intervention immediately. The follow-up questionnaire to measure at 3 months and 6 months after intervention.
  Seven statements were used to assessment the attitude toward oral care, including' oral cleansing is a part of elderly people daily body cleaning.' A score was used the Liker scale with rating from 1 (completely disagree) to 5 (completely agree) was used for each statement. The total score ranged was 7-35.
Self-efficacy of oral care | After randomization, HCWs would receive pre-test before intervention and post-test after intervention immediately. The follow-up questionnaire to measure at 3 months and 6 months after intervention.
  Nine statements were used to measures the self-efficacy to oral care , including 'I am confident in helping elderly people brush their teeth with the modified Bass brushing technique.' A score was used the Liker scale with rating from 1 (completely disagree) to 5 (completely agree) was used for each statement. The total score was 9-45.
Intention to assist in oral care behavior | After randomization, HCWs would receive pre-test before intervention and post-test after intervention immediately.
  Eight statements were used to evaluate the intention to assist in oral care behavior , including 'I will take the initiative to assist the elderly in using the modified Bass brushing technique to brush their teeth.' A score was used the Liker scale with rating from 1 (completely disagree) to 5 (completely agree) was used for each statement. The total score ranged was 8-40.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Ling Huang, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Sanmin Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No